CLINICAL TRIAL: NCT00831649
Title: A Phase II, Multicenter, Open-Label, Long-Term Study of the Safety, Tolerability, and Efficacy of Intravenous Natalizumab in Subjects With Rheumatoid Arthritis Who Have Previously Participated in Study ELN100226-RA201
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The biological effect seen with natalizumab was not sufficient to warrant further development in RA.
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELN100226-RA251
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2009-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Natalizumab

ARMS (1):
- natalizumab (Experimental)
  Interventions: Drug: natalizumab

INTERVENTIONS:
Drug: natalizumab
  Other Names: TYSABRI

SUMMARY:
The purpose of this study is to evaluate the long-term safety, tolerability, and efficacy of natalizumab in subjects with active rheumatoid arthritis (RA) receiving concomitant methotrexate (MTX)

ELIGIBILITY:
INCLUSION CRITERIA

Subjects will be eligible to begin study participation if they meet all of the following inclusion criteria:

* Subjects must give written informed consent
* Male or female subjects ≥18 to ≤75 years of age (at randomization in Study ELN100226-RA201)
* Subjects must have been randomized in Study ELN100226-RA201;
* Subjects who have completed the Month 6 visit of Study ELN100226-RA201 OR Subjects who have an inadequate therapeutic response (defined as a < 20% reduction from baseline [Month 0 in Study ELN100226-RA201] for both painful/tender and swollen joint counts) after receiving at least 4 infusions of study drug and has not been rescued with other RA medications during the treatment phase of Study ELN100226-RA201;
* Subjects must be taking MTX at the same dose last used in Study ELN100226-RA201;
* Female subjects of childbearing potential agreed to use adequate, contraceptive methods (either intrauterine device [IUD], oral or depot contraceptive, or barrier plus spermicide). Female subjects of childbearing potential used adequate contraception for at least 2 months prior to study entry and continued contraception for at least 3 months after their last infusion of study drug;
* Subjects must be willing and able to complete all planned study procedures.

EXCLUSION CRITERIA

Subjects will be excluded from the study if they meet any of the following exclusion criteria:

* Females who are pregnant or breastfeeding or those planning to become pregnant in the next 14 months;
* Subjects who have experienced anaphylaxis, angioedema, urticaria, clinical syndrome diagnostic of serum sickness, or biopsy-proven vasculitis to a previous infusion of study drug;
* Subjects who received rescue intervention in Study ELN100226-RA201, defined as an increase in dose of an existing permitted concomitant treatment of RA or the introduction of a new treatment of RA;
* Subject who are expected to be unavailable for the duration of the trial, likely to be noncompliant with the Protocol, or who are felt to be unsuitable by the Investigator for any other reason;
* Subjects with a history of a malignancy (other than surgically excised basal or squamous cell carcinoma of the skin);
* Subjects with a history of clinically significant and/or persistent gastrointestinal, pulmonary, chronic infection, cardiovascular, renal, hepatic, neurological, dermatological, immunological, major psychiatric (including drug or alcohol abusers) or hematological illness, which in the opinion of the Investigator places the subject at unacceptable risk for participation in the study;
* Subjects who intend to donate blood or blood products during the period of the study or within one month following completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-09; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
The number and proportion of subjects with AEs
The number and proportion of subjects with SAEs
The number and percentage of subjects who discontinue early from the study due to an AE
Assessment of clinical laboratory parameters, physical examination, and vital signs.